CLINICAL TRIAL: NCT03950141
Title: Apatinib Combined With S-1 as Maintenance Therapy for HER-2 Negatived Gastric Cancer Treated With 4 Cycles Chemotherapy Valued as Stable Disease (SD)
Brief Title: Apatinib Combined With S-1 as Maintenance Therapy for HER-2 Negatived Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yingying Huang, Principal Investigator, Beijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017BJYYH-053-02
Record Dates: First submitted 2018-11-18; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: HER-2 Negatived Gastric Cancer
MeSH Terms: interventions — apatinib; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib and S1 group (Experimental): Combined with Apatinib (250mg qd po) and S-1 (40-60mg bid d1-14) as maintenance therapy in advanced HER-2 negatived GC
  Interventions: Drug: Apatinib and S-1

INTERVENTIONS:
Drug: Apatinib and S-1 — Combined with Apatinib (250mg qd po) and S-1 (40-60mg bid d1-14) as maintenance therapy in advanced HER-2 negatived GC

SUMMARY:
Apatinib is a novel drug which was produced by Jiangsu Hengrui Medicine Co.Ltd in China. It is approved in advanced gastric cancer（GC）. The investigators just want to design such kind of trail to prove its effect when combined with S-1 as maintenance in advanced HER-2 negatived GC treated with 4 cycles chemotherapy and valued as SD. Investigators will evaluate progression free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
GC is the second most common cause of cancer-related deaths worldwide. Most patients are diagnosed with unresectable advanced or metastatic stage disease losing the radical surgery opportunity. Till now there is no novel targeted drug which can increase the OS for advanced GC patients except HER-2 positive patients.

Approximate 30 patients with unresectable GC treated with 4 cycles chemotherapy and valued as stable disease will be enrolled in this study,The investigators will evaluate the efficacy and security of apatinib and S-1 as maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proved advanced HER-2 negatived gastric adenocarcinoma;
2. At least a unresectable factor before operation via CT, MRI, or PET-CT: difficult resection of locally advanced gastric cancer(T4b); hepatic metastasis (H1; at most five lesions, total diameter ≤8 cm); Peritoneal metastasis(CY1, P1) ; Definitely diagnosed as unresectable GC via exploratory laparoscopy or laparotomy;
3. ECOG performance status 0-2;
4. Age≥ 18 years old, Life expectancy estimated than 3 months;
5. For results of blood routine test and biochemical tests:

   Hgb ≥ 80g/L, WBC ≥ 4000/mm3, ANC ≥ 1.5×109/L, platelets ≥ 80×109/L ALT and AST ≤ 2.5 x upper normal limit (UNL), and ≤ 5 x UNL（Hematogenous metastases）, Serum Total bilirubin ≤ 1.5 X UNL, Serum Creatine ≤ 1.5 x UNL ；
6. Good cardiac function before the recruitment, no seizure of myocardial infarction in past half years, and controllable hypertension and other coronary heart disease;
7. Not concomitant with other uncontrollable benign disease before the recruitment(e.g. the infection in the kidney, lung and liver);
8. Informed consent.

Exclusion Criteria:

1. Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management;
2. Coronary heart disease greater than Class I; I-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class I cardiac dysfunction;
3. Patients with positive urinary protein;
4. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
5. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 2 months;
6. Contraindications include allergy to apatinib and/or its accessories, active bleeding, intestinal perforation, intestinal obstruction, within 30 days after surgery, drugs with poor-controlled hypertension, Class Ⅲ-Ⅳ cardiac dysfunction （NYHA standard）, severe hepatic and renal dysfunction（level 4）if apatinib use is considered;
7. Abnormal Coagulation (INR>1.5, APTT>1.5 UNL), with tendency of bleed;
8. Pregnant or lactating women; Any other condition that might place the patient at undue risk or preclude a patient from completing the study;
9. Treated with 4 cycles chemotherapy included Tegafur;
10. Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | Patients will be followed for an average period of 1 year
  From date of registration until the date of disease progresssion or death resulting from any cause.

SECONDARY OUTCOMES:
overall survival | Patients will be followed for an average period of 1 year
  From date of registration until the date of death from any cause or the last follow-up visit.

OTHER OUTCOMES:
1-year survival rate | 12 months
  Percentage of patients alive at 1 year.
Safety and tolerability as measured by number and grade of toxicity events | 12 months
  Overall Safety Profile by CTCAE V4.1

CONTACTS AND LOCATIONS:
Overall Officials: yingying Huang, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No